CLINICAL TRIAL: NCT02144376
Title: Validation of Magnetic Resonance Imaging to Characterise Gastrointestinal Physiology, Gut Luminal Content and Its Interaction With Colonic Microbiota in Patients With Chronic Constipation
Brief Title: MRI and Microbiota Analysis in Constipation
Acronym: MIMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UON14011; 14GA006 (Other: Nottingham University Hospitals NHS Trust)
Record Dates: First submitted 2014-03-25; First posted 2014-05-22 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Constipation
Keywords: Constipation; psyllium; ispaghula; Magnetic Resonance Imaging; MRI; microbiota
MeSH Terms: conditions — Constipation | interventions — Psyllium; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Placebo Comparator): 7 days without use of laxatives other than standardised rescue therapy 7 grams maltodextrin taken 3 times daily, at least 4 hours apart, for up to 7 days
  Interventions: Dietary Supplement: Maltodextrin
- Ispaghula (Active Comparator): 7 days without use of laxatives other than standardised rescue therapy 7 grams ispaghula/ psyllium taken 3 times daily, at least 4 hours apart, for up to 7 days
  Interventions: Dietary Supplement: Ispaghula

INTERVENTIONS:
Dietary Supplement: Ispaghula
  Other Names: psyllium
  Arms: Ispaghula
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
The purpose of the study is to test how well magnetic resonance imaging (MRI) can measure whole gut transit time in people with constipation, and how readily it can detect a change in transit time induced by taking a dietary supplement with laxative effects.The investigators expect to demonstrate that ispaghula (psyllium) accelerates movement of matter through the intestinal tract.

The investigators will also assess whether a change in gut bacteria and the chemicals that they release can be detected.

ELIGIBILITY:
Inclusion Criteria:

* Meets Rome III Criteria for diagnosis of Functional Constipation5 on questionnaire (NB. Both those who do and do not meet IBS criteria will be eligible)
* At least one bowel motion per week while taking usual laxatives
* Able to give informed consent
* Aged 18 or older

Exclusion Criteria:

* History declared by the candidate of other pre-existing gastrointestinal disorder, including but not limited to:
* Inflammatory Bowel Disease
* Coeliac Disease diagnosed in the last year
* Pancreatitis
* Cancer of the gastrointestinal tract
* Any reported history of gastrointestinal resection (excluding appendicectomy or cholecystectomy)
* Presence of an intestinal stoma
* Pregnancy declared by candidate (no formal testing)
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Reported alcohol intake of >28 units/ week with daily drinking
* Any use of a product containing ispaghula or psyllium in the 4 weeks prior to consent
* Unable to avoid use of dihydrocodeine or morphine during the study
* If taking other regular opiates such as codeine, fentanyl or Oxycodone, participants should be able to maintain a stable dose throughout the study
* Any reported history of hypersensitivity or significant adverse reaction to ispaghula, maltodextrin or bisacodyl
* Unable to stop drugs and other agents used primarily for their laxative effect, during periods of screening, washout, baseline and treatment (maximum 15 days - rescue medication will be provided).
* Antibiotic or prescribed probiotic treatment in the past 4 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in any medical trials for the past 3 months
* Any condition where the candidate is likely to require a course of antibiotics in the next 3 months e.g. severe chronic respiratory disease, recurrent urinary tract infection, lower limb ulceration
* Judgement by the PI that the candidate who will be unable to comply with the full study protocol e.g. Diabetes, severe COPD

During the screening 2 weeks off laxatives

* No bowel motions recorded during screening period
* ≥3 complete spontaneous bowel motions (CSBMs - bowel motion with the feeling of complete evacuation, without the use of rescue therapy in the preceding 24 hours) per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Weighted Average Position Score of transit marker capsules as determined by MRI | 24 hours after ingestion
  After 4 days of study product participants will ingest 5 transit mark capsules, the use of which has been shown to measure whole gut transit in a similar manner to more established techniques. They will continue to take study product before undergoing an MRI scan to assess capsule position

SECONDARY OUTCOMES:
Weighted Average Position Score of 5 transit marker capsules, as determined by MRI | 48 hours after ingestion
  After 4 days of study product participants will ingest 5 transit mark capsules, the use of which has been shown to measure whole gut transit in a similar manner to more established techniques. They will continue to take study product before undergoing an MRI scan to assess capsule position
Small Bowel Water Content (SBWC) in millilitres(mL) measured by MRI | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve (mL.min) will be calculated from hourly MRI scans
Small Bowel Water Content (SBWC) in millilitres measured by MRI | Baseline, 60 minutes before test meal
  After 5 days of taking the study product participants will undergo an MRI scan while fasted.
Ascending Colon Water Content in millilitres measured by MRI | Baseline, 60 minutes before test meal
  After 5 days taking study product participants will undergo an MRI scan while fasted
Ascending Colon Water Content in millilitres measured by MRI | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve (mL.min) will be calculated from hourly MRI scans
Change from baseline in Ascending Colon Water Content in millilitre measured by MRI | test meal -60, test meal +60
  Difference between measurement Meal -60 (fasting) and Meal +60
Change from before to after challenge meal in Ascending Colon Water Content before in millilitre measured by MRI | test meal +360 minutes, test meal + 420 minutes
  Difference between time points Meal2 -20 and Meal 2 +40
Ascending Colon T1 | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve of MRI parameter measured at hourly time points
Descending Colon T1 | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve of MRI parameter measured at hourly time points
Ascending colon T2 | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve of MRI parameter measured at hourly time points
Descending Colon T2 | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve of MRI parameter measured at hourly time points

OTHER OUTCOMES:
Colonic volume | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve (mL.min) will be measured from hourly MRI scans by segmentation into ascending colon (AC), transverse colon (TC) and descending colon (DC)
Colonic gas volume | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve (mL.min), measured on hourly MRI scans by segmentation into AC, TC and DC
Gastric volume | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Area under the curve (mL.min) measured on hourly MRI scans
Abdominal circumference | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  Measured at the umbilicus in cm, determined by MRI
Change from baseline of stool water content percentage by mass | after an average 5 days of intervention
  Stool will be sampled during the baseline week and between days 3-7 of the intervention week during each treatment period
Change from baseline in stool frequency | during days 9-14 of treatment period
  Each treatment period includes 1 day washout, 7 days baseline, up to 7 (minimum 6) days intervention. Total = 15 days.
  Stool frequency will be sampled on days 2-8 and 9-14, since participants may stop taking intervention before day 15.
Change from baseline in stool consistency | During days 9-14 of treatment period
  Each treatment period includes 1 day washout, 7 days baseline, up to 7 (minimum 6) days intervention. Total = 15 days.
  Stool consistency will be sampled on days 2-8 and 9-14, since participants may stop taking intervention before day 15.
Change from baseline in faecal microbiota | Change from baseline after an average 5 days of intervention
  Will be assessed for relative abundance, richness and diversity
Change from baseline in faecal short-chain fatty acids | Change from baseline after an average 5 days of intervention
  Stool samples collected during baseline week and after 3 or more days of intervention in each treatment period.
Symptoms during study day | -60, 0, 60, 120, 180, 240, 300, 360, 420 minutes after test meal
  4 symptoms will be measured on 2 scales: a previously validated questionnaire on an ordinal scale (OS) of 0 (none), 1 (mild/ distinct but negligible), 2 (moderate/ annoying), 3 (severe/ disabling); and a Visual Analogue Scale (VAS) (0-100)
  Symptoms include abdominal pain, bloating, gas/flatulence, and diarrhoea. Clinically important symptoms will be defined as additive total score of 3 or greater on OS. VAS scores will be analysed alongside MRI data

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MSc MD FRCP, Study Chair — University of Nottingham; Giles Major, BM BCh MRCP, Principal Investigator — University of Nottingham; Luca Marciani, MSc PhD, Study Director — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No